CLINICAL TRIAL: NCT04429698
Title: The Effects of Point-of-care Ultrasonography on the Dıagnosıs Process of Patıents Who Admıtted to Emergency Department: Randomised-Controlled Trial
Brief Title: The Effects of Point-of-care Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Necip Gökhan Güner, Principial Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 05 of 12.09.2018
Record Dates: First submitted 2020-06-05; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Chest Pain
Keywords: chest pain, POCUS, length of stay, emergency department
MeSH Terms: conditions — Chest Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POCUS group (Other): Patients in this group underwent POCUS after primary clinical evaluation with the knowledge of their primary physician. This procedure was performed in the first hour after the patients' primary clinical evaluations to evaluate the predetermined parameters in the study form for the heart, lungs, hepatobiliary, aortic and deep veins.
  Interventions: Diagnostic Test: Point of care ultrasonography
- Control group (No Intervention): All processes and results were followed without any intervention in the processes related to the patients in this group and the results were recorded in the study form

INTERVENTIONS:
Diagnostic Test: Point of care ultrasonography — Point-of-care Ultrasonography is an imaging method performed with ultrasound aid to facilitate rapid diagnosis and interventions during emergency intervention.
  Arms: POCUS group

SUMMARY:
Background: When used with standard diagnostic testing, point-of-care ultrasonography (POCUS) might improve the proportion of patients admitted with chest pain (CP) who are correctly diagnosed, decrease length of stay (LOS) in emergency department (ED) and costs. We therefore assessed POCUS for the heart, lungs, aortic, hepatobiliary and deep vein in addition to the usual initial diagnostic testing in this patient population.

Methods: In a prospective, randomised-controlled, parallel-group trial in the ED at Sakarya University Training and Research Hospital, Turkey, patients (≥18 years) with CP were randomly assigned in a 1:1 ratio to a standard diagnostic strategy (control group) or to standard diagnostic strategy supplemented with POCUS (POCUS group).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency were included in this study if they had chest pain, or chest pain with back pain, neck and jaw pain, abdominal pain, arm pain and shortness of breath

Exclusion Criteria:

* permanent mental disability
* age younger than 18 years
* having chest trauma in the last 24 hours
* to be pregnant
* need for urgent angiography with ST elevation myocardial infarction
* to be referred to the ED as a diagnosis of external center
* failure to obtain complete patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization or discharge | 6 months
Average costs during the diagnosis of patients. | 6 months

SECONDARY OUTCOMES:
The rate of change in the preliminary diagnosis of physician | 6 months
The Hospitalization rate | 6 months
The discharge rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Necip G Guner, M.D., Principal Investigator — Sakarya University Training and Research Hospital
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buhumaid RE, St-Cyr Bourque J, Shokoohi H, Ma IWY, Longacre M, Liteplo AS. Integrating point-of-care ultrasound in the ED evaluation of patients presenting with chest pain and shortness of breath. Am J Emerg Med. 2019 Feb;37(2):298-303. doi: 10.1016/j.ajem.2018.10.059. Epub 2018 Oct 30. PMID 30413369
- [Result] Laursen CB, Sloth E, Lassen AT, Christensen Rd, Lambrechtsen J, Madsen PH, Henriksen DP, Davidsen JR, Rasmussen F. Point-of-care ultrasonography in patients admitted with respiratory symptoms: a single-blind, randomised controlled trial. Lancet Respir Med. 2014 Aug;2(8):638-46. doi: 10.1016/S2213-2600(14)70135-3. Epub 2014 Jul 3. PMID 24998674
- [Result] Lamsam L, Gharahbaghian L, Lobo V. Point-of-care Ultrasonography for Detecting the Etiology of Unexplained Acute Respiratory and Chest Complaints in the Emergency Department: A Prospective Analysis. Cureus. 2018 Aug 28;10(8):e3218. doi: 10.7759/cureus.3218. PMID 30405993
- [Result] Elikashvili I, Tay ET, Tsung JW. The effect of point-of-care ultrasonography on emergency department length of stay and computed tomography utilization in children with suspected appendicitis. Acad Emerg Med. 2014 Feb;21(2):163-70. doi: 10.1111/acem.12319. PMID 24673672
- [Result] Lin MJ, Neuman M, Rempell R, Monuteaux M, Levy J. Point-of-Care Ultrasound is Associated With Decreased Length of Stay in Children Presenting to the Emergency Department With Soft Tissue Infection. J Emerg Med. 2018 Jan;54(1):96-101. doi: 10.1016/j.jemermed.2017.09.017. Epub 2017 Oct 27. PMID 29110982